CLINICAL TRIAL: NCT02507323
Title: TIPRIS: Ticagrelor vs. Prasugrel Effects on Infarct Size: A Head to Head Comparison With Prasugrel
Brief Title: Ticagrelor vs. Prasugrel Effects on Infarct Size
Acronym: TIPRIS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: collaborator withdrew the study
Sponsor: Yochai Birnbaum (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Yochai Birnbaum, Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 34665: Ticagrelor v Prasugrel
Record Dates: First submitted 2015-07-17; First posted 2015-07-23 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ticagrelor or matching placebo (Active Comparator): ticagrelor (180 mg loading followed by 90 mg twice daily) or matching placebo
  Interventions: Drug: ticagrelor; Drug: Placebo
- prasugrel or matching placebo (Active Comparator): prasugrel (60 mg loading followed by 5-10 mg/d) or matching placebo
  Interventions: Drug: prasugrel; Drug: Placebo

INTERVENTIONS:
Drug: ticagrelor — A platelet aggregation inhibitor
  Other Names: Brilinta
  Arms: ticagrelor or matching placebo
Drug: prasugrel — a thienopyridine class inhibitor of platelet activation and aggregation
  Other Names: Effient
  Arms: prasugrel or matching placebo
Drug: Placebo — placebo

SUMMARY:
This study has been designed as a randomized, double-blind trial to provide definitive evidence on the effects of ticagrelor and prasugrel on myocardial salvage in patients with anterior ST Segment Elevation Myocardial Infarction (STEMI) undergoing primary Percutaneous Coronary Intervention (PCI). This study will also measure the effects of ticagrelor vs. prasugrel on secondary endpoints listed above. This study design aims to test the hypothesis that ticagrelor will reduce myocardial infarct size as a proportion of the ischemic area at risk when compared to prasugrel.

DETAILED DESCRIPTION:
Subjects and research staff (including the Magnetic Resonance Imaging (MRI) readers and interventional cardiologists) will not know what active treatment study drug the subjects are receiving.

Study Arm 1: Ticagrelor (180 mg loading dose, followed by 90 mg twice a day) PO plus matching placebo

Study Arm 2: Prasugrel (60 mg loading dose followed by 5 or 10 mg once per day based on weight) PO plus matching placebo

Additional study drug: Aspirin (81mg per day)

Participation in this study will be about 90 days and includes 4 study visits (other than your hospital stay) and 3 telephone calls.

ENROLLMENT PROCEDURES:

The following procedures are to be completed after informed consent has been obtained:

* Informed Consent Form signed
* Medical history
* Vital signs (eg, blood pressure, heart rate, respiration rate, temperature)
* Review for Adverse Events (AEs) and Serious Adverse Events (SAEs) (only AEs possibly related to study procedures and SAEs are collected)
* Documentation of concomitant medications
* Physical exam
* Body height
* Body weight
* 12-lead Electrocardiogram (ECG)
* Angiographic and Percutaneous Coronary Intervention (PCI) data
* Randomization of treatment assignment
* Investigational product dispensing (on Day 0 and during hospital stay) - Loading dose on Day 0 - 3 day investigational product dosing while in the hospital - 30 day supply dispensing of investigational product on Day 3 for subject to take home
* Local laboratory Assessments: - Blood draw for Creatine Kinase-MB (CK-MB) and troponin I - Blood pregnancy (females of childbearing potential only)

FOLLOW UP PROCEDURES:

Day 5

* Vital signs (e.g., blood pressure, heart rate, respiration rate, temperature)
* Review for Adverse Events and Serious Adverse Events (only AEs possibly related to study procedures and SAEs are collected)
* Cardiac MRI
* Left Ventricular Ejection Fraction (LVEF), Left Ventricular End-Diastolic Volume (LVEDV), Left Ventricular End-Systolic Volume (LVESV) calculations
* Serum creatinine, Complete Blood Count (CBC)
* Documentation of concomitant medications and investigational product compliance

Day 30 (+/- 1 day), Day 60 (+/- 2 days)

* Vital signs (e.g., blood pressure, heart rate, respiration rate, temperature)
* Review for Adverse Events and Serious Adverse Events (only AEs possibly related to study procedures and SAEs are collected)
* LVEF, LVEDV, LVESV calculations
* Serum creatinine, CBC
* Documentation of concomitant medications and investigational product compliance
* Investigational Product Dispensing

Day 14, Day 44, Day 74 (+/- 2 days):

Phone calls will be performed to ensure drug compliance, review concomitant medications and review any events. On Day 74, study staff will confirm whether or not the subject has seen their regular cardiologist. Subject will be instructed to bring this information with them at the Day 90 visit so that their cardiologist can be told what arm they participated in for continuation of care and medication therapy.

Day 90 or Termination/End of Study (+/- 2 days) :

* Vital signs (eg, sitting blood pressure, heart rate, respiration rate, temperature)
* Review for Adverse Events and Serious Adverse Events (only AEs possibly related to study procedures and SAEs are collected)
* Cardiac MRI
* LVEF, LVEDV, LVESV calculations
* Serum creatinine, CBC
* Documentation of concomitant medications and investigational product compliance
* If available and subject consents, subject's cardiologist will be informed what arm of the study they participated in for continuation of care and medication therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: Signed informed consent prior to any study specific procedures
2. Age: Male and females aged 18 years and older
3. Onset: Presenting to emergency room or cardiac catheterization laboratory within 6 hours of onset of myocardial infarction symptoms
4. Continuing to have ongoing myocardial infarction symptoms
5. EKG findings: ST elevation on ECG with positive T waves in the precordial leads, suggestive of anterior STEMI
6. Triaged for emergency cardiac catheterization (primary PCI protocol)
7. Agree to use an effective contraceptive method beginning at the signing of the informed consent and for at least 30 days after the last dose of study drug. The definition of an effective method of contraception will be based on the judgment of the investigator.

Exclusion Criteria:

1. Prior myocardial infarction
2. Contraindication to ticagrelor and/or prasugrel
3. Contraindication to gadolinium
4. Contraindication to aspirin
5. Treatment with fibrinolytic therapy for the index STEMI
6. High risk of bleeding
7. Presenting with cardiogenic shock
8. Infarction due to stent thrombosis
9. History of a previous coronary artery bypass graft (CABG)
10. Known renal insufficiency (acute kidney injury or Glomerular Filtration Rate < 40 mL/min/1.73 m2).
11. Moderate or severe hepatic impairment
12. Inability to undergo cardiac MRI
13. Indication for aspirin >162 mg/d
14. Indication for Nonsteroidal Anti-Inflammatory Drugs or COX2 inhibitors
15. Pregnant
16. Breast feeding
17. History of intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy as measured by infarct size on all randomized patients. | up to Day 90

SECONDARY OUTCOMES:
Safety as measured by incidences of treatment emergent adverse events, serious adverse events, treatment-related adverse events and adverse events leading to stop of drug | 90 days
  for 90 day major adverse cardiac events and bleeding complications

CONTACTS AND LOCATIONS:
Overall Officials: Yochai Birnbaum, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Baylor-St. Lukes Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas